CLINICAL TRIAL: NCT06081530
Title: Single-blind, Randomised, Placebo-Controlled Trial on the Safety, Tolerability, and Pharmacokinetics of Single Rising Doses and Multiple Doses of Intravenous BI 3802876 in Healthy Subjects
Brief Title: A Study in Healthy Men to Test How Well Different Doses of BI 3802876 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1517-0001; 2023-504538-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-06; First posted 2023-10-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part A: BI 3802876 dose group 1 (Experimental)
  Interventions: Drug: BI 3802876
- Part A: BI 3802876 dose group 2 (Experimental)
  Interventions: Drug: BI 3802876
- Part A: BI 3802876 dose group 3 (Experimental)
  Interventions: Drug: BI 3802876
- Part A: BI 3802876 dose group 4 (Experimental)
  Interventions: Drug: BI 3802876
- Part A: BI 3802876 dose group 5 (Experimental)
  Interventions: Drug: BI 3802876
- Part A: BI 3802876 dose group 6 (Experimental)
  Interventions: Drug: BI 3802876
- Part A: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3802876
- Part B: BI 3802876 (Experimental)
  Interventions: Drug: BI 3802876
- Part B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3802876

INTERVENTIONS:
Drug: BI 3802876 — BI 3802876
  Arms: Part A: BI 3802876 dose group 1; Part A: BI 3802876 dose group 2; Part A: BI 3802876 dose group 3; Part A: BI 3802876 dose group 4; Part A: BI 3802876 dose group 5; Part A: BI 3802876 dose group 6; Part B: BI 3802876
Drug: Placebo matching BI 3802876 — Placebo matching BI 3802876
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The main objective of this trial is to investigate the safety, tolerability, and pharmacokinetics of BI 3802876 when administered in different doses in healthy male volunteers. The primary objective is to descriptively assess the frequency of drug-related adverse events (AEs) in subjects treated with BI 3802876, as compared to placebo. The secondary objective is to descriptively assess pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (temperature, blood pressure, pulse), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of ≥18 to ≤55 years at screening
3. Body mass index (BMI) of ≥ 19.0 to ≤ 28.0 kg/m2 at screening. A minimum body weight of 65 kg at screening
4. Signed and dated written informed consent prior to admission to the study, in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) and local legislation

Exclusion Criteria:

1. Any finding in the medical examination (including blood pressure (BP), pulse rate, or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Three repeated measurements of systolic BP outside the range of 80 to 130 mm Hg, diastolic BP outside the range of 50 to 80 millimetre of mercury (mmHg), or pulse outside the range of 45 to 90 beats per minute.
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator

Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Occurrences of any drug-related AEs between first drug administration (BI 3802876 or placebo) and end of the residual effect period (REP) | up to Day 35 for Part A and up to Day 117 for Part B

SECONDARY OUTCOMES:
Part A: Area under the concentration-time curve of the analyte in serum over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to Day 35
Part A: Maximum measured concentration of the analyte in serum (Cmax) | up to Day 35
Part B: Area under the concentration-time curve of the analyte in serum over the dosing interval tau at steady state, if steady state can be reasonably assumed (AUCτ,ss) | up to Day 117
Part B: Maximum measured concentration of the analyte in serum at steady state, if steady state can be reasonably assumed (Cmax,ss) | up to Day 117

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com